CLINICAL TRIAL: NCT00114231
Title: A Phase II Trial of Chemoradiotherapy and Local Excision for uT2uN0 Rectal Cancer
Brief Title: Capecitabine, Oxaliplatin, and Radiation Therapy in Treating Patients Who Are Undergoing Surgery for Stage I Rectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACOSOG-Z6041; ACOSOG-Z6041; U10CA180821 (NIH); U10CA076001 (NIH); CDR0000433145 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2005-06-13; First posted 2005-06-14 (Estimated); Results first posted 2018-03-29 (Actual); Last update posted 2018-03-29 (Actual); Status verified 2018-02

CONDITIONS: Colorectal Cancer
Keywords: adenocarcinoma of the rectum; stage I rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Rectal Neoplasms | interventions — Capecitabine; Oxaliplatin; Neoadjuvant Therapy; Radiotherapy; Radiation; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (capecitabine, oxaliplatin, radiotherapy, surgery) (Experimental): Patients undergo high-dose external beam radiotherapy once daily and receive capecitabine PO BID on days 1-5, 8-12, 15-19, 22-26, and 29-33. Patients also receive oxaliplatin IV over 2 hours on days 1, 8, 22, and 29.
  Approximately 4-8 weeks after completion of chemoradiotherapy, patients undergo local excision of the tumor. Patients with T3 disease or positive resection margins after local excision undergo radical resection of the rectum and receive additional chemotherapy and/or radiotherapy at the discretion of the physician.
  Interventions: Drug: capecitabine; Drug: oxaliplatin; Procedure: neoadjuvant therapy; Radiation: radiation therapy

INTERVENTIONS:
Drug: capecitabine
  Other Names: Given IV
Drug: oxaliplatin — Given IV
Procedure: neoadjuvant therapy — Undergo surgery
  Other Names: therapeutic conventional surgery
Radiation: radiation therapy — Undergo radiotherapy
  Other Names: irradiation, radiotherapy, therapy, radiation

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as capecitabine and oxaliplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Oxaliplatin may make tumor cells more sensitive to radiation therapy. Giving capecitabine and oxaliplatin together with radiation therapy before surgery may shrink the tumor so it can be removed.

PURPOSE: This phase II trial is studying how well giving capecitabine and oxaliplatin together with radiation therapy works in treating patients who are undergoing surgery for stage I rectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the 3-year disease-free survival rate in patients with stage I adenocarcinoma of the rectum treated with neoadjuvant chemoradiotherapy comprising capecitabine, oxaliplatin, and radiotherapy followed by local excision.

Secondary

* Determine the rate of resectability with negative resection margins in patients treated with this regimen.
* Determine the procedure-specific morbidity and mortality in patients treated with this regimen.
* Determine the rate of pathologic complete response of the primary tumor in patients treated with this regimen.
* Determine the impact of this regimen on anorectal function and quality of life in these patients.
* Determine the feasibility of using molecular studies to assess surgical resection margins and tumor response in patients treated with this regimen.
* Determine molecular markers associated with local tumor recurrence in patients treated with this regimen.

OUTLINE: This is a non-randomized, multicenter study.

Patients undergo high-dose external beam radiotherapy once daily on days 1-5, 8-12, 15-19, 22-26, and 29-33. Patients also receive oral capecitabine twice daily on days 1-14 and 22-35 and oxaliplatin IV over 2 hours on days 1, 8, 22, and 29. Approximately 4-8 weeks after completion of chemoradiotherapy, patients undergo local excision of the tumor. Patients with T3 disease or positive resection margins after local excision undergo radical resection of the rectum and receive additional chemotherapy and/or radiotherapy at the discretion of the physician.

Quality of life is assessed at baseline and then 1 year after surgery.

After completion of study treatment, patients are followed at 1 month, every 4 months for 3 years, and then every 6 months for 2 years.

PROJECTED ACCRUAL: A total of 102 patients will be accrued for this study within 2.8 years.

ELIGIBILITY:
* Patient must have an Eastern Cooperative Oncology Group (ECOG)/Zubrod status of =< 2
* Patient must have histologically confirmed invasive adenocarcinoma of the rectum; Note: patients with rectal tumors suspicious for invasion also are eligible
* Distal border of the patient's tumor must be within 8 cm from the anal verge as measured on endoscopic exam
* Patients with tumors fixed to adjacent structures on digital exam are NOT eligible
* Patient must have an uT2uN0 tumor, as confirmed by endorectal ultrasound (ERUS) or endorectal coil magnetic resonance imaging (MRI) scan; patients with uT1, uT3, or uT4 tumors are NOT eligible; greatest diameter of tumor cannot exceed 4 cm
* Patients with positive perirectal nodes on ERUS examination are NOT eligible
* Patients with histologic evidence of metastatic invasion of inguinal lymph nodes are NOT eligible
* Patients with the following conditions are NOT allowed on study:

  * Metastatic disease or other primaries (patient must have had chest X-ray/computed tomography [CT] and abdominal & pelvic CT/MRI with IV contrast, as well as a colonoscopy)
  * Previously documented history of familial adenomatous polyposis
  * Previously documented history of hereditary non-polyposis colorectal cancer diagnosed clinically (Amsterdam II criteria) or by genetic testing
  * History of inflammatory bowel disease
  * History of prior radiation treatments to pelvis
  * Clinically significant peripheral sensory or motor neuropathy (defined as symptomatic weakness, paresthesia or sensory alteration described to be interfering with function, interfering with activities of daily living, disabling or life-threatening)
  * History of any clinically significant cardiac disease (i.e., class 3-4 congestive heart failure, symptomatic coronary artery disease, uncontrolled arrhythmia, and/or myocardial infarction within the last 6 months)
  * History of uncontrolled seizures or clinically significant central nervous system disorders
  * History of psychiatric conditions or diminished mental capacity that could compromise the giving of informed consent, or interfere with study compliance
  * History of allergy and/or hypersensitivity to capecitabine and/or oxaliplatin
  * History of difficulty or inability to take or absorb oral medications
* White blood cells (WBC) >= 3000/mm^3
* Absolute neutrophil count (ANC) > 1,500/mm^3
* Hemoglobin > 9.5 mg/dl
* Platelet count >= 100,000/mm^3
* Total bilirubin =< 3 mg/dl
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.0 times institutional upper limit of normal (ULN)
* Alkaline phosphatase =< 2.0 times ULN
* Creatinine clearance (CLcr) >= 50 ml/min by Cockroft-Gault equation
* Patients who have experienced a prior malignancy must have received potentially curative therapy for that malignancy, and must be cancer-free for at least five years from the date of initial diagnosis (exceptions: patients treated for non-melanoma skin carcinoma, or in-situ carcinomas)
* Patients of reproductive potential must agree to use an effective method of birth control when undergoing treatments with known or possible mutagenic or teratogenic effects; all female participants of childbearing potential must have a negative urine or serum pregnancy test within two weeks prior to study registration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2006-05; Primary Completion 2013-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julio Garcia-Aguilar, MD, PhD, Study Chair — City of Hope Comprehensive Cancer Center
Locations (67):
- United States (67):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Cancer Care Center at John Muir Health - Concord Campus, Concord, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Chao Family Comprehensive Cancer Center at University of California Irvine Medical Center, Orange, California
  - John Muir/Mt. Diablo Comprehensive Cancer Center, Walnut Creek, California
  - St. Vincent's Medical Center, Bridgeport, Connecticut
  - Praxair Cancer Center at Danbury Hospital, Danbury, Connecticut
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Tampa General Hospital, Tampa, Florida
  - Curtis and Elizabeth Anderson Cancer Institute at Memorial Health University Medical Center, Savannah, Georgia
  - Nancy N. and J. C. Lewis Cancer and Research Pavilion at St. Joseph's/Candler, Savannah, Georgia
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - William N. Wishard Memorial Hospital, Indianapolis, Indiana
  - Reid Hospital & Health Care Services, Richmond, Indiana
  - Ochsner Cancer Institute at Ochsner Clinic Foundation, New Orleans, Louisiana
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Altru Cancer Center at Altru Hospital, Grand Forks, North Dakota
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Clinton Memorial Hospital, Wilmington, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Integris Oncology Services, Oklahoma City, Oklahoma
  - Natalie Warren Bryant Cancer Center at St. Francis Hospital, Tulsa, Oklahoma
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - Knight Cancer Institute at Oregon Health and Science University, Portland, Oregon
  - Morgan Cancer Center at Lehigh Valley Hospital - Cedar Crest, Allentown, Pennsylvania
  - UPMC Cancer Center at Beaver Medical Center, Beaver, Pennsylvania
  - UPMC Cancer Center at Jefferson Regional Medical Center, Clairton, Pennsylvania
  - UPMC Cancer Center - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - UPMC Cancer Center at the John P. Murtha Pavilion, Johnstown, Pennsylvania
  - UPMC - Moon, Moon Township, Pennsylvania
  - UPMC Cancer Center - Natrona Heights, Natrona Heights, Pennsylvania
  - Jameson Memorial Hospital - North Campus, New Castle, Pennsylvania
  - Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania
  - Allegheny Cancer Center at Allegheny General Hospital, Pittsburgh, Pennsylvania
  - UPMC - Shadyside, Pittsburgh, Pennsylvania
  - UPMC Cancer Center at Magee-Womens Hospital, Pittsburgh, Pennsylvania
  - UPMC Cancer Center at UPMC Presbyterian, Pittsburgh, Pennsylvania
  - UPMC Cancer Center at UPMC St. Margaret, Pittsburgh, Pennsylvania
  - Western Pennsylvania Cancer Institute at Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - UPMC Cancer Centers, Pittsburgh, Pennsylvania
  - UPMC Cancer Center at UPMC Passavant, Pittsburgh, Pennsylvania
  - St. Clair Memorial Hospital Cancer Center, Pittsburgh, Pennsylvania
  - UPMC Cancer Center at UPMC Northwest, Seneca, Pennsylvania
  - Washington Hospital Cancer Center, Washington, Pennsylvania
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - M. D. Anderson Cancer Center at University of Texas, Houston, Texas
  - Methodist Hospital, Houston, Texas
  - Surgical Oncology Associates, Newport News, Virginia
  - Providence Cancer Center at Sacred Heart Medical Center, Spokane, Washington
  - Providence Cancer Center at Holy Family Hospital, Spokane, Washington
  - United Hospital Center, Clarksburg, West Virginia
  - Edwards Comprehensive Cancer Center at Cabell Huntington Hospital, Huntington, West Virginia
  - University of Wisconsin Paul P. Carbone Comprehensive Cancer Center, Madison, Wisconsin

REFERENCES:
- [Background] Ota DM, Nelson H; ACOSOG Group Co-Chairs. Local excision of rectal cancer revisited: ACOSOG protocol Z6041. Ann Surg Oncol. 2007 Feb;14(2):271. doi: 10.1245/s10434-006-9213-7. Epub 2006 Nov 14. No abstract available. PMID 17103255
- [Result] Garcia-Aguilar J, Shi Q, Thomas CR Jr, Chan E, Cataldo P, Marcet J, Medich D, Pigazzi A, Oommen S, Posner MC. A phase II trial of neoadjuvant chemoradiation and local excision for T2N0 rectal cancer: preliminary results of the ACOSOG Z6041 trial. Ann Surg Oncol. 2012 Feb;19(2):384-91. doi: 10.1245/s10434-011-1933-7. Epub 2011 Jul 14. PMID 21755378
- [Result] Garcia-Aguilar J, Renfro LA, Chow OS, Shi Q, Carrero XW, Lynn PB, Thomas CR Jr, Chan E, Cataldo PA, Marcet JE, Medich DS, Johnson CS, Oommen SC, Wolff BG, Pigazzi A, McNevin SM, Pons RK, Bleday R. Organ preservation for clinical T2N0 distal rectal cancer using neoadjuvant chemoradiotherapy and local excision (ACOSOG Z6041): results of an open-label, single-arm, multi-institutional, phase 2 trial. Lancet Oncol. 2015 Nov;16(15):1537-1546. doi: 10.1016/S1470-2045(15)00215-6. Epub 2015 Oct 22. PMID 26474521

RESULTS

PARTICIPANT FLOW:
Groups:
- Original Dose Group: External beam radiotherapy with megavoltage linear accelerators (≥ 6 MV) was delivered to a 3-4 field pelvis arrangement after CT-based simulation and computer-assisted treatment planning. Intensity-modulated radiotherapy was allowed. The original dose of radiotherapy was 1·8 Gy per day, 5 days a week for 5 weeks to a dose of 45 Gy to planning target volume 1, then a boost of 9 Gy to planning target volume 2 (defi ned as the gross tumour volume plus 2 cm) for a total dose of 54 Gy. This was accompanied by capecitabine (825 mg/m², twice daily, on days 1-14 and 22-35) and oxaliplatin (50 mg/m² on weeks 1, 2, 4, and 5). Surgery was done 4-8 weeks after completion of neoadjuvant chemoradiotherapy. Local excision was done using conventional transanal excision or transanal endoscopic microsurgery. Full-thickness excision of the tumour with a 1 cm surrounding margin of normal rectal wall was needed.
- Revised Dose Group: The radiotherapy was reduced to a total of 50·4 Gy by reducing the 9 Gy boost to 5·4 Gy, and capecitabine was reduced to 725 mg/m², twice daily, 5 days a week for 5 weeks. The dose of oxaliplatin was not changed. Surgery was done 4-8 weeks after completion of neoadjuvant chemoradiotherapy. Local excision was done using conventional transanal excision or transanal endoscopic microsurgery. Full-thickness excision of the tumour with a 1 cm surrounding margin of normal rectal wall was needed.
Period: Overall Study
Arm/Group | Original Dose Group | Revised Dose Group
Started | 62 | 28
Completed | 53 | 26
Not Completed | 9 | 2
Not completed — No consent | 2 | 0
Not completed — QARC requirement not met | 1 | 0
Not completed — Suspected metastatic disease | 1 | 0
Not completed — No adenocarcinoma | 1 | 0
Not completed — Low creatinine clearance | 0 | 1
Not completed — Tumor size > 4cm | 1 | 0
Not completed — Tumor fixed on digital exam | 0 | 1
Not completed — No Absolute Neutrophil Count | 2 | 0
Not completed — Biopsy done after registration | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Original Dose Group | Revised Dose Group | Total
Number analyzed (Participants) | 53 | 26 | 79
Age, Continuous [Median (Full Range); unit: years] | 62 [30 to 80] | 63 [45 to 83] | 62 [30 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 6 | 26
  Male | 33 | 20 | 53
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 53 | 26 | 79

OUTCOME MEASURES:

1. Primary Outcome: 3-Year Disease-free Survival
Description: The primary endpoint was 3-year disease-free survival (DFS). Evidence of local recurrence, distant metastasis, or death from any cause within 3 years counted as events in the time-to-event Kaplan-Meier analysis of disease-free survival.
Time Frame: Up to 3 years
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Treatment (Capecitabine, Oxaliplatin, Radiotherapy, Surgery)
Number analyzed (Participants) | 79
percentage of patients | 88.2 [81.3 to 95.8]

2. Secondary Outcome: R0 Resection Rate (Negative Margin Rate)
Description: The rate (percentage) of patients with negative resection margins after undergoing local excision is reported below.
Time Frame: At time of surgery
Population: Patients who had local excision are included in this analysis.
Measure: Number; unit: percentage of patients
Arm/Group | Treatment (Capecitabine, Oxaliplatin, Radiotherapy, Surgery)
Number analyzed (Participants) | 77
percentage of patients | 98.7

3. Secondary Outcome: Morbidity and Mortality Rate
Description: Morbidity and mortality after neoadjuvant cheoradiotherapy and local excision.
Time Frame: Up to 30 days
Measure: Number; unit: percentage of patients
Arm/Group | Treatment (Capecitabine, Oxaliplatin, Radiotherapy, Surgery)
Number analyzed (Participants) | 79
percentage of patients
  Mortality | 6
  Morbidity | 10

4. Secondary Outcome: Rate of Pathologic Complete Response of the Primary Tumor
Description: The rate (percentage) of patients with pathologic complete response (pCR) is reported below. Pathologic response will be determined by comparing tumor width and stage in the surgical specimen with the same parameters as determined by pre-CRT ERUS: PATHOLOGIC COMPLETE RESPONSE (pCR): no residual tumor.
Time Frame: Up to 5 years
Population: Patients assessable for pathology results were included in this analysis.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Treatment (Capecitabine, Oxaliplatin, Radiotherapy, Surgery)
Number analyzed (Participants) | 77
percentage of patients | 44 [32 to 55]

5. Secondary Outcome: Local Recurrence Rate
Description: The local recurrence rate (percentage) is defined as the percentage of patients who had local recurrence as initial sites of failure at the end of follow-up.
Time Frame: Up to 5 years
Measure: Number; unit: percentage of patients
Arm/Group | Treatment (Capecitabine, Oxaliplatin, Radiotherapy, Surgery)
Number analyzed (Participants) | 79
percentage of patients | 4

ADVERSE EVENTS:
Time Frame: Up to 3 years.
Description: Each CTCAE term is a unique representation of a specific event used for medical documentation and scientific analysis and is a single MedDRA Lowest Level Term (LLT). All graded AEs are reported for those who received at least one dose of CRT. Serious AE (SAE) reports may include any secondary serious or non-serious events considered related to the primary event (the reason for filing an expedited report); collectively, these events are referred to as Expedited AEs, and appear in the SAE table.
Arm/Group | Original Dose Group | Revised Dose Group
All-Cause Mortality (participants affected / at risk) | 0/57 | 0/27
Serious Adverse Events (participants affected / at risk) | 6/57 | 2/27
Other Adverse Events (participants affected / at risk) | 32/57 | 25/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Original Dose Group (N=57) | Revised Dose Group (N=27)
Hemoglobin decreased (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Myocardial ischemia (Cardiac disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Serum phosphate decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Serum potassium decreased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hematoma (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Original Dose Group (N=57) | Revised Dose Group (N=27)
Blood disorder (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hemoglobin decreased (Blood and lymphatic system disorders) | 3 (8) | 13 (40)
Lymphatic disorder (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Myocardial ischemia (Cardiac disorders) | 1 (2) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Diplopia (Eye disorders) | 0 (0) | 1 (3)
Vision blurred (Eye disorders) | 0 (0) | 4 (8)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 7 (10)
Anal exam abnormal (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anal pain (Gastrointestinal disorders) | 0 (0) | 3 (3)
Anal ulcer (Gastrointestinal disorders) | 1 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 9 (15)
Diarrhea (Gastrointestinal disorders) | 20 (35) | 21 (73)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 0 (0) | 1 (1)
Endoscopy small intestine abnormal (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enteritis (Gastrointestinal disorders) | 0 (0) | 2 (5)
Fecal incontinence (Gastrointestinal disorders) | 0 (0) | 3 (5)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 4 (7)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 8 (10) | 15 (30)
Proctitis (Gastrointestinal disorders) | 0 (0) | 2 (5)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (3)
Rectal pain (Gastrointestinal disorders) | 6 (9) | 13 (39)
Rectal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (5) | 4 (6)
Chills (General disorders) | 0 (0) | 3 (3)
Edema limbs (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 7 (14) | 18 (60)
Fever (General disorders) | 1 (1) | 3 (3)
Flu-like symptoms (General disorders) | 0 (0) | 1 (1)
Localized edema (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 4 (7) | 5 (6)
Infection (Infections and infestations) | 2 (2) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Radiation recall reaction (dermatologic) (Injury, poisoning and procedural complications) | 6 (8) | 7 (16)
Rectal anastomotic leak (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 4 (4)
Bilirubin increased (Investigations) | 0 (0) | 3 (5)
Creatinine increased (Investigations) | 0 (0) | 1 (2)
INR increased (Investigations) | 0 (0) | 2 (3)
Laboratory test abnormal (Investigations) | 0 (0) | 1 (1)
Leukocyte count decreased (Investigations) | 1 (1) | 8 (30)
Lymphocyte count decreased (Investigations) | 2 (4) | 9 (29)
Neutrophil count decreased (Investigations) | 0 (0) | 5 (13)
Platelet count decreased (Investigations) | 1 (2) | 5 (20)
Serum cholesterol increased (Investigations) | 0 (0) | 1 (1)
Weight loss (Investigations) | 1 (2) | 5 (11)
Anorexia (Metabolism and nutrition disorders) | 3 (4) | 10 (20)
Blood glucose increased (Metabolism and nutrition disorders) | 3 (9) | 9 (28)
Blood uric acid increased (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Dehydration (Metabolism and nutrition disorders) | 3 (5) | 4 (4)
Serum albumin decreased (Metabolism and nutrition disorders) | 0 (0) | 5 (11)
Serum calcium decreased (Metabolism and nutrition disorders) | 0 (0) | 4 (5)
Serum calcium increased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Serum potassium decreased (Metabolism and nutrition disorders) | 1 (2) | 3 (6)
Serum potassium increased (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Serum sodium decreased (Metabolism and nutrition disorders) | 1 (1) | 6 (8)
Serum sodium increased (Metabolism and nutrition disorders) | 1 (3) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 2 (3)
Neurological disorder NOS (Nervous system disorders) | 1 (3) | 2 (6)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 2 (4)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (3) | 7 (13)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Taste alteration (Nervous system disorders) | 0 (0) | 4 (9)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (2)
Depression (Psychiatric disorders) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 2 (9)
Libido decreased (Psychiatric disorders) | 0 (0) | 1 (1)
Bladder spasm (Renal and urinary disorders) | 0 (0) | 1 (1)
Cystitis (Renal and urinary disorders) | 0 (0) | 1 (1)
Glomerular filtration rate decreased (Renal and urinary disorders) | 0 (0) | 1 (6)
Urethral pain (Renal and urinary disorders) | 0 (0) | 3 (7)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 9 (20)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Urogenital disorder (Renal and urinary disorders) | 1 (2) | 1 (2)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 3 (3)
Perineal pain (Reproductive system and breast disorders) | 0 (0) | 2 (3)
Testicular pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1)
Hemorrhage nasal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (4)
Rash desquamating (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (3)
Sweating (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Hot flashes (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 3 (4)
Hypotension (Vascular disorders) | 1 (1) | 1 (1)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes